CLINICAL TRIAL: NCT03394898
Title: Prospective, Observational Study of Evaluation of Body Mass Index and Eating Behaviour Changes in Female Patients With Fibromyalgia Under Medical Treatment
Brief Title: Evaluation of Body Mass Index and Eating Behaviour Changes in Female Patients With Fibromyalgia Under Medical Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Alper Mengi, Alper Mengi, M.D., Gaziosmanpasa Research and Education Hospital
Other Study IDs: 27.12.2017/108
Record Dates: First submitted 2018-01-03; First posted 2018-01-09 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Eating Behavior; Body Weight; Fibromyalgia
Keywords: Chronic Pain; Body Mass Index; Eating Habits
MeSH Terms: conditions — Feeding Behavior; Body Weight; Fibromyalgia; Chronic Pain | interventions — Body Mass Index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: body mass index, eating behaviour — The patients' weights and heights will be measured and the body mass index will be calculated from the measured values.Patients' eating behaviour will be questioned with Three Factor Eating Questionnaire. The 18-item Three-Factor Eating Questionnaire is a scale that measures three domains of eating behavior: cognitive restraint , uncontrolled eating and emotional eating.

SUMMARY:
The purpose of this study is to evaluate of body mass index and eating behaviour changes in female patients with fibromyalgia under medical treatment.

DETAILED DESCRIPTION:
The female patients with fibromyalgia under medical treatment say that body mass index and eating behaviour changes,for this reason, this relationship will be investigated in this study.

Demographic data (sex, age, education level, occupation) of patients with fibromyalgia diagnosis will be questioned and height lengths will be measured. The group of medications (serotonin and norepinephrine reuptake inhibitor or GABAergic drugs) that begins with the diagnosis of the disease fibromyalgia will be recorded.

All patients will be assessed when diagnosed, followed by 2nd week and then 4nd week.

In each follow-up, the patients' weights will be measured again (the body mass index will be calculated from the measured value).

In each follow-up, the effect of fibromyalgia on the daily life of the patients will be questioned with Fibromyalgia Impact Questionnaire (FIQ). The FIQ was developed from information gathered from patient reports, functional status instruments, and clinical observations. This instrument measures physical functioning, work status (missed days of work and job difficulty), depression, anxiety, morning tiredness, pain, stiffness, fatigue, and well-being over the past week.

In each follow-up, patients' eating behaviour will be questioned with Three Factor Eating Questionnaire. The 18-item Three-Factor Eating Questionnaire is a scale that measures three domains of eating behavior: cognitive restraint , uncontrolled eating and emotional eating.

In each follow-up, the right calf circumference of the patients will be measured in centimeters with a tape measure .

ELIGIBILITY:
Inclusion Criteria:

* Female subjects between the ages of 18-40
* Subjects, who met the 2013 American College of Rheumatology (ACR) criteria for Fibromyalgia

Exclusion Criteria:

* History of eating disorders such as anorexia nervosa, bulimia nevroza
* History of hypothyroidism or hyperthyroidism
* Pregnant or breast feeding
* History of central or peripheral nervous system disorders
* History of infectious, chronic inflammatory disease, malignant tumors
* Subjects with active psychiatric illness or who use psychiatric medication
* Uncooperative subject
* History of cardiac pathology such as heart failure, coronary artery disease
* History of diabetes, chronic renal insufficiency, chronic liver failure

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Being a female between the ages of 18-40
Study Population: Subjects who applied to the Physical Medicine and Rehabilitation outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01-03 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
eating behaviour | 7 days
  Patients' eating behaviour will be questioned with Three Factor Eating Questionnaire. The 18-item Three-Factor Eating Questionnaire is a scale that measures three domains of eating behavior: cognitive restraint , uncontrolled eating and emotional eating.

SECONDARY OUTCOMES:
activities of daily living | 7 days
  The effect of fibromyalgia on the daily life of the patients will be questioned with Fibromyalgia Impact Questionnaire (FIQ). The FIQ was developed from information gathered from patient reports, functional status instruments, and clinical observations. This instrument measures physical functioning, work status (missed days of work and job difficulty), depression, anxiety, morning tiredness, pain, stiffness, fatigue, and well-being over the past week.
calf circumference | 1 day
  The right calf circumference of the patients will be measured in centimeters with a tape measure .
body mass index | 1 day
  The patients' weights and heights will be measured and the body mass index will be calculated from the measured values.

CONTACTS AND LOCATIONS:
Overall Officials: alper MENGİ, M.D., Principal Investigator — Gaziosmanpasa Taksim Training and Research Hospital
Locations (1):
- Gaziosmanpasa Taksim Research and Education Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim CH, Luedtke CA, Vincent A, Thompson JM, Oh TH. Association of body mass index with symptom severity and quality of life in patients with fibromyalgia. Arthritis Care Res (Hoboken). 2012 Feb;64(2):222-8. doi: 10.1002/acr.20653. PMID 21972124